CLINICAL TRIAL: NCT01166503
Title: Early Versus Delayed Surgery for Infantile Esotropia: A Clinical Evaluation of Sensory and Motor Outcomes
Brief Title: Early Versus Delayed Surgery for Infantile Esotropia
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Agnes Wong, Ophthamologist-In-Chief, The Hospital for Sick Children
Other Study IDs: 1000005134
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Esotropia
Keywords: pediatrics; Esotropia; Surgery
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Surgery: This group will be made up of subjects whose parents choose to have them undergo corrective surgery at or before age 11 months.
  Interventions: Procedure: mVEP Testing; Procedure: Stereoacuity Testing; Procedure: Optokinetic nystagmus testing; Procedure: Motion detection testing; Procedure: Motion discrimination testing
- Standard Surgery: This group will be made up of subjects who present after age 11 months or whose parents choose to have them undergo corrective surgery between 11-18 months.
  Interventions: Procedure: mVEP Testing; Procedure: Stereoacuity Testing; Procedure: Optokinetic nystagmus testing; Procedure: Motion detection testing; Procedure: Motion discrimination testing

INTERVENTIONS:
Procedure: mVEP Testing — Five small sensors are placed on the head which record the brain's response to moving stripes that are displayed on a computer screen. Each eye is tested while the other eye is patched. Each recording trial lasts about 10 seconds, and several trials are done for each eye.
Procedure: Stereoacuity Testing — Subjects will have their 3D perception measured using standard clinical stereo tests (Randot, Lang, Titmus).
Procedure: Optokinetic nystagmus testing — Subjects will be asked to view a screen with vertical stripes moving in both leftward and rightward directions while their eye movements are recorded using a remote video-based eye tracker.
Procedure: Motion detection testing — Subjects will view a computer screen that has two panels of dots on them. The subject will be required to pick which panel has a section of dots that are moving in a specific direction (ie. nasalward/temporalward).
Procedure: Motion discrimination testing — Subjects will view a computer screen that has two panels of randomly moving dots on them. The subject will be required to pick which panel has a section of dots that are moving in a specific direction (ie. nasalward/temporalward).

SUMMARY:
The goal of this study is to determine whether corrective surgery done earlier than the current standard can better improve the visual and eye movement deficits in children with infantile esotropia (crossed eyes in infancy).

DETAILED DESCRIPTION:
While there is a uniform agreement among pediatric ophthalmologists that most infantile esotropia requires surgical correction, the proper timing of surgery is controversial. In North America, the typical age at surgery ranges from 11-18 months. Unfortunately, despite successful surgical realignment of the eyes, the sensory and eye movement deficits often persist. Recently, some pediatric ophthalmologists have advocated earlier surgery. The rationale for early surgery stems from animal and human research showing that early realignment of the eyes within an early critical period allows normal development of the sensory and eye movement systems.

ELIGIBILITY:
Inclusion Criteria:

1. onset of esotropia after 10 weeks of age;
2. constant esotropia ≥ 20° (40 prism diopter or PD) at near (1/3 m) on two examinations, separated by 2-4 weeks; and
3. refractive error ≤ +3.00 diopters (far-sightedness).

Exclusion Criteria:

1. gestational age < 34 weeks;
2. birth weight ≤ 1500 g;
3. ventilator treatment in the newborn period;
4. history of meningitis or other major medical event;
5. developmental delay;
6. incomitant or paralytic strabismus;
7. manifest nystagmus or head bobbing;
8. prior eye muscle surgery;
9. prior treatment of amblyopia or spectacle correction for refractive errors;
10. presence of structural ocular anomalies.

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with infantile esotropia will be enrolled from The Hospital for Sick Children in Toronto. Infants with characteristics that indicate low likelihood of spontaneous resolution will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2004-05; Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Motion visual evoked potential (mVEPs) asymmetry | at age 2 years
  mVEP measures the perception of nasalward and temporalward motion for each eye at the cortical level. A nasal bias index (NBI) is calculated, which will show whether subjects perceive motion better for one direction over the other.
Stereopsis | at 2 and 5 years of age
  This measures the level of 3D depth perception.
Optokinetic nystagmus (OKN) asymmetry | at age 5 years
  OKN is measured in both the nasalward and temporalward directions for each eye. From this a nasal bias index (NBI) is calculated, which will show whether subjects perceive motion better in one direction or the other.
Global Motion Perception | at 2 and 5 years of age
  Motion perception will be tested using two tasks: motion detection (at age 2 and 5 years) and motion discrimination (at age 5 years).

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Wong, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No